CLINICAL TRIAL: NCT00149253
Title: A Randomized, Double-Blind, Controlled Trial of Etoricoxib as a Pre-Emptive Analgesic for Abdominal Hysterectomy
Brief Title: Pre-Emptive Analgesia Efficacy of Etoricoxib for Postoperative Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: acute pain service; Faculty of Medicine,KhonKaenU
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2005-09-08 (Estimated); Status verified 2004-10

CONDITIONS: a Single-Dose of Etoricoxib; Post-Operative Morphine Consumption; Total Pain Relief Over 8 Hr(TOPAR8); Post Transabdominal Hysterectomy
Keywords: Abdominal hysterectomy,; Etoricoxib,; morphine consumption,; pre-emptive analgesia

INTERVENTIONS:
Drug: a single-dose of Etoricoxib before induction of anesthesia

SUMMARY:
Taken together, studies of the value of pre-emptive analgesia are inconclusive. This randomized, double-blind, dose-ranging, placebo-controlled study was therefore designed to test that a reduction in post-operative morphine consumption can be achieved by a single-dose of etoricoxib before induction of anesthesia.

DETAILED DESCRIPTION:
Patients undergoing transabdominal hysterectomy were randomized to a group taking a single dose (orally) of etoricoxib 120 mg (n = 18), etoricoxib 180 mg (n = 17) or placebo (n = 15) 2 hours before surgery under the same standardized general anesthesia. At the post-anesthetic care unit, intravenous morphine titration was given before starting self-controlled analgesia (PCA) device. Morphine consumption, pain relief score, sedative score, global evaluation score, and side-effects were recorded at 1, 2, 4, 8 and 24 h post-operatively. The primary end points were morphine consumption within 24-hr post-operatively and total pain relief over 8 h (TOPAR8). Patient global satisfaction was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* The ASA I or II patients undergoing elective transabdominal hysterectomy with general anesthesia

Exclusion Criteria:

* Patients with history of opioid addiction or chronic pain
* Allergy to other nonsteroidal anti-inflammatory, or asthma
* Concomitant use of tricyclic antidepressants, opioid analgesics, antihistamines, tranquilizers, hypnotics, sedatives, or systemic corticosteroids
* Those unable to understand the principle of patient-controlled analgesia(PCA) device were excluded from the study

Ages: 15 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2004-12; Study Completion 2005-05

PRIMARY OUTCOMES:
The primary end points were morphine consumption within 24-hr post-operatively
and total pain relief over 8 h (TOPAR8).

SECONDARY OUTCOMES:
Patient global response to therapy

CONTACTS AND LOCATIONS:
Overall Officials: waraporn chau-in, Asso Prof., Principal Investigator — Department of Anesthesiology, Faculty of Medicine,KhonKaen University,KhonKaen 40002, Thailand
Locations (1):
- Warporn Chau-in, KhonKaen University, KhonKaen, Thailand